CLINICAL TRIAL: NCT03234556
Title: Diagnosing Clinically Significant Prostate Cancer in African American and White Men Phase II, Randomized Clinical Trial, Multi-center, MR-Guided vs. 12-core Systematic Random Biopsy, Localized Prostate Cancer
Brief Title: Diagnosing Clinically Significant Prostate Cancer In African American and White Men With Elevated PSA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 4P-16-7; NCI-2017-00890 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 4P-16-7 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH); R01CA205058 (NIH)
Record Dates: First submitted 2017-07-26; First posted 2017-07-31 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Health Status Unknown; Elevated PSA
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Arm I (SR-Bx) (Active Comparator): Patients undergo SR-Bx. If SR-Bx doesn't reveal clinically significant cancer, then MRI will be done in 3 months, and if lesion is present (PIRADS ≥ 3) schedule for MRUS-Bx. If there is no lesion, then no biopsy. Schedule MRI in 12 months after the initial MRI.
  Interventions: Procedure: Biopsy of Prostate; Other: Laboratory Biomarker Analysis; Diagnostic Test: Magnetic Resonance Imaging; Diagnostic Test: MRI Ultrasound Fusion Guided Biopsy
- Arm II (MRI, MRUS-Bx, SR-Bx) (Experimental): Patients undergo MRI. Must be scheduled at least one day before MRUS biopsy.
  * If MRI shows no lesion present (PIRADS 1-2), then no MRUS-Bx. Schedule for SR-Bx only.
  * If MRI shows lesion present (PIRADS ≥ 3), perform MRUS-Bx, which will be done first and followed immediately by SR-Bx.
  Interventions: Procedure: Biopsy of Prostate; Other: Laboratory Biomarker Analysis; Diagnostic Test: Magnetic Resonance Imaging; Diagnostic Test: MRI Ultrasound Fusion Guided Biopsy

INTERVENTIONS:
Procedure: Biopsy of Prostate — Undergo SR-Bx
  Other Names: Prostate Biopsy; Prostatic Biopsy
Other: Laboratory Biomarker Analysis — Correlative studies
Diagnostic Test: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Diagnostic Test: MRI Ultrasound Fusion Guided Biopsy — Undergo MRUS-Bx
  Other Names: Fusion Biopsy; Fusion-Guided Biopsy; MR Fusion Biopsy; MRI-Ultrasound Fusion Biopsy; MRI/Ultrasound Fusion Biopsy; MRI/US Biopsy

SUMMARY:
This randomized phase II trial studies how well systematic random biopsy or magnetic resonance imaging (MRI)-ultrasound image (US) fusion biopsy work in diagnosing prostate cancer in patients with elevated prostate specific antigen. Systematic random biopsy and MRI-US fusion biopsy may work better in improving the accuracy of prostate cancer detection.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the detection of clinically significant prostate cancer (CSPCa) in Arm 1 versus Arm 2.

II. To compare between African American (AA) and white men the probability of developing CSPCa within three years of initial biopsy at the start of the study.

SECONDARY OBJECTIVES:

I. To determine complications and patient morbidity associated with either systematic random prostate biopsy (SR-Bx) versus (vs) magnetic resonance imaging-ultrasound image fusion biopsy (MRUS-Bx) + SR-Bx.

TERTIARY OBJECTIVES:

I. To compare Gleason score between MRUS-Bx and radical prostatectomy (RP) specimen among men who elect RP (~110 in the randomized controlled trial [RCT]).

II. To assess within Arm 1 the detection of CSPCa three months after SR-Bx among men initially diagnosed with clinically insignificant prostate cancer (CinsPCa) or no cancer.

III. To identify among men invited to participate and those actually enrolled in the RCT: determinants of study participation.

IV. To identify among men invited to participate and those actually enrolled in the RCT: determinants of treatment decision (active surveillance [AS] vs radiation vs RP) including the diagnostic method.

OUTLINE: Patients are randomized into 1 of 2 arms.

ARM I: SR-Bx group

* Patients undergo SR-Bx

  * If SR-Bx doesn't reveal clinically significant cancer, then MRI in 3 months, and if lesion is present (PIRADS ≥ 3) schedule for MRUS-Bx.
  * If there is no lesion, then no biopsy - schedule MRI in 12 months after the initial MRI.

ARM II: MRUS-Bx group

* Patients undergo MRI. Must be scheduled at least 1 day before MRUS Biopsy.

  * MRI shows no lesion present (PIRADS 1-2): no MRUS-Bx, schedule for SR-Bx only.
  * MRI lesion present (PIRADS ≥ 3): schedule for MRUS-Bx, which will be done first and followed immediately after by SR-Bx.

FOLLOW UP:

After completion of procedure, patients are followed up at 2-4 weeks, 3, 6, 9, and 12 months, and then periodically for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization for release of personal health information

  * Note: HIPAA authorization may be included in the informed consent or obtained separately
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 1 within 3 months (93 days) prior to being registered for protocol
* African-American or white men (Hispanic or non-Hispanic)
* Prostate biopsy-naive or a single negative biopsy
* Having elevated prostate specific antigen (PSA) (> 2.5 ng/ml) and no palpable nodule on digital rectal exam (DRE)
* Ability to understand the willingness to sign a written informed consent
* Patients must be willing to undergo a radiologic imaging before and after biopsy of the prostate
* Patients must be willing to undergo a biopsy of the prostate

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 12 months of the study for other diagnoses not related to prostate cancer
* Patients receiving any other investigational agents
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with active inflammatory bowel disease
* Patients who are unable to undergo MRI
* Patients who had any surgery of the prostate including TURP (transurethral resection of the prostate)
* Patients who had > 1 prior prostate biopsy

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-05-23 (Estimated)

PRIMARY OUTCOMES:
Biopsy detection rate of clinically significant prostate cancer | Up to 5 years
  Will code patients as having clinically significant prostate cancer if they are diagnosed with Gleason score >= 7 or any Gleason score with core length >= 5 mm or any Gleason score that includes Gleason pattern >= 4 at initial systematic random biopsy.

SECONDARY OUTCOMES:
Presence of any of the complications | Up to 5 years
  Will be summarized in the complications checklist. Will determine any striking co-morbidities that are present post-biopsy and were absent pre-biopsy within each arm, and next determine if the prevalence of any of these identified post-biopsy morbidities differs between the two arms. For these analyses, regression methods (linear, logistic, multinomial logistic as appropriate for the "dependent" variable being analyzed) will be used. Standard descriptive methods will be used to summarize and display the results.

OTHER OUTCOMES:
Highest Gleason score | Up to 5 years
  Will assess the highest Gleason score in magnetic resonance imaging-ultrasound image fusion biopsy and systematic random biopsy. Will evaluated using agreement metrics such as percent agreement, Cohen's kappa (k) statistic and Krippendorff's alpha statistic. Significance will be considered if p < 0.05.

CONTACTS AND LOCATIONS:
Overall Officials: Inderbir Gill, Principal Investigator — University of Southern California
Locations (4):
- United States (4):
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of Maryland, Baltimore, Maryland
  - Henry Ford Hospital Vattikuti Urology Institute, Detroit, Michigan
  - Memorial Sloan-Kettering Cancer Center, New York, New York